CLINICAL TRIAL: NCT02868385
Title: Repeated Doses of Praziquantel in Schistosomiasis Treatment (RePST): An Open Label, Randomized Controlled Trial of Single vs. Multiple Treatments of Praziquantel in Intestinal African Schistosomiasis in Côte d'Ivoire
Brief Title: Repeated Doses of Praziquantel in Schistosomiasis Treatment (RePST)
Acronym: RePST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Swiss Tropical & Public Health Institute (Other); Centre Suisse de Recherches Scientifiques en Cote d'Ivoire (Other)
Responsible Party: Principal Investigator, Meta Roestenberg, MD PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RePST; 2016-003017-10 (EudraCT Number)
Record Dates: First submitted 2016-08-09; First posted 2016-08-16 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Schistosomiasis
Keywords: Schistosomiasis; Schistosoma mansoni; Bilharzia
MeSH Terms: conditions — Schistosomiasis | interventions — Praziquantel

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (A) (Active Comparator): 1x praziquantel: Children assigned to group A receive a standard single oral dose of praziquantel (40 mg/kg) at baseline (week 0) and will receive no further treatment until the final visit (week 8).
  Interventions: Drug: 1x Praziquantel
- Intervention group (B) (Experimental): 4x praziquantel: Children assigned to group B receive a standard single oral dose of praziquantel (40 mg/kg) at baseline (week 0) and will receive three consecutive praziquantel treatments (40 mg/kg) in the following six weeks with 2 weeks intervals.
  Interventions: Drug: 4x Praziquantel

INTERVENTIONS:
Drug: 4x Praziquantel — Four consecutive praziquantel treatments (40 mg/kg): at baseline (week 0) and at week 2, 4, and 6.
  Other Names: Biltricide
  Arms: Intervention group (B)
Drug: 1x Praziquantel — One praziquantel treatment (40 mg/kg) at baseline
  Other Names: Biltricide
  Arms: Control group (A)

SUMMARY:
An open label, randomized controlled trial of single vs. multiple treatments of praziquantel in intestinal African schistosomiasis in Côte d'Ivoire

This study aims to determine the efficacy of repeated (up to four times) praziquantel treatment against S. mansoni infection in school-age children from Côte d'Ivoire using the traditional Kato-Katz thick smear technique, but also with more accurate and non-invasive antigen- and DNA-detection methods.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a confirmed S. mansoni infection (positive POC-CCA test result and at least one positive out of triplicate Kato-Katz thick smears)
* Subject is aged between 5 and 18 years and otherwise in good health
* Subject has received no recent praziquantel treatment in the past month
* Subject has provided oral assent and provided written informed consent signed by parents/legal guardian
* Subject is able and willing to provide multiple stool and urine samples during study

Exclusion Criteria:

* Known allergy to study medication (i.e. praziquantel and albendazole)
* Pregnancy
* Lactating

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 167 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Cure rate | 8 weeks
  The difference in cure rate (percentage negative) between intervention and control arm by Kato-Katz technique

SECONDARY OUTCOMES:
Reduction rates | 8 weeks
  The difference in egg reduction rate (by Kato-Katz), cure rate and circulating anodic and cathodic antigen and DNA reduction rate after multiple doses of praziquantel (40 mg/kg) by Kato Katz (KK), point-of-care circulating cathodic antigen assay (POC-CCA), up-converting phosphor lateral flow circulating anodic antigen assay (UCP-LF-CAA) and polymerase chain reaction (PCR), respectively.
Sensitivity and specificity | 8 weeks
  Sensitivity and specificity of Kato Katz (KK), point-of-care circulating cathodic antigen assay (POC-CCA), up-converting phosphor lateral flow circulating anodic antigen assay (UCP-LF-CAA) and polymerase chain reaction (PCR) at different time points.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Coulibaly, Principal Investigator — Centre Suisse de Recherches Scientifiques en Cote d'Ivoire
Locations (1):
- Centre Suisse de Recherches Scientifiques en Côte d'Ivoire, Abidjan, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoekstra PT, Casacuberta Partal M, Amoah AS, van Lieshout L, Corstjens PLAM, Tsonaka S, Assare RK, Silue KD, Meite A, N'Goran EK, N'Gbesso YK, Roestenberg M, Knopp S, Utzinger J, Coulibaly JT, van Dam GJ. Repeated doses of Praziquantel in Schistosomiasis Treatment (RePST) - single versus multiple praziquantel treatments in school-aged children in Cote d'Ivoire: a study protocol for an open-label, randomised controlled trial. BMC Infect Dis. 2018 Dec 14;18(1):662. doi: 10.1186/s12879-018-3554-2. PMID 30547750
- [Result] Hoekstra PT, Casacuberta-Partal M, van Lieshout L, Corstjens PLAM, Tsonaka R, Assare RK, Silue KD, Meite A, N'Goran EK, N'Gbesso YK, Amoah AS, Roestenberg M, Knopp S, Utzinger J, Coulibaly JT, van Dam GJ. Efficacy of single versus four repeated doses of praziquantel against Schistosoma mansoni infection in school-aged children from Cote d'Ivoire based on Kato-Katz and POC-CCA: An open-label, randomised controlled trial (RePST). PLoS Negl Trop Dis. 2020 Mar 20;14(3):e0008189. doi: 10.1371/journal.pntd.0008189. eCollection 2020 Mar. PMID 32196506
- [Derived] Hoekstra PT, Casacuberta-Partal M, van Lieshout L, Corstjens PLAM, Tsonaka R, Assare RK, Silue KD, N'Goran EK, N'Gbesso YK, Brienen EAT, Roestenberg M, Knopp S, Utzinger J, Coulibaly JT, van Dam GJ. Limited efficacy of repeated praziquantel treatment in Schistosoma mansoni infections as revealed by highly accurate diagnostics, PCR and UCP-LF CAA (RePST trial). PLoS Negl Trop Dis. 2022 Dec 22;16(12):e0011008. doi: 10.1371/journal.pntd.0011008. eCollection 2022 Dec. PMID 36548444